CLINICAL TRIAL: NCT02320955
Title: Swiss Prospective Autologous Bone Flap Resorption Study
Acronym: SPARS
Status: Terminated | Type: Observational
Why Stopped: Interim analysis confirmed too high rate of bone flap resorption. Continuation of the study was deemed unethical. Available data allow evaluation with sufficient power.
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ZH-2014-0370
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Brain Edema
Keywords: autologous bone flap; decompressive craniectomy; malignant brain swelling; patient specific implant; bone resorption; aseptic bone necrosis
MeSH Terms: conditions — Brain Edema; Bone Resorption; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reimplantation of cryoconserved bone flap: All patients who receive reimplantation of a cryoconserved autologous bone flap
  Interventions: Procedure: Reimplantation of cryoconserved bone flap

INTERVENTIONS:
Procedure: Reimplantation of cryoconserved bone flap — A bone flap, which was explanted for decompression of a swollen brain or following severe head trauma and which was cryoconserved in the meantime is reimplanted. This procedure is the gold-standard therapy after decompressive hemicraniectomy and is routinely performed.

SUMMARY:
The complications after reimplantation of cryoconserved autologous bone flaps are reported inhomogeniously in the literature. Especially the incidence of bone flap resorption varies from 0% to about 30%. More recent retrospective studies seem to find higher resorption rates and thus suggest to implant artificial bone replacements from the start. The Swiss Prospective Autologous bone Resorption Study is the first propspective observational study designed to determine the true incidence of autologous bone resorption.

DETAILED DESCRIPTION:
Patients undergoing decompressive craniectomy and delayed reimplantation of the cryoconserved autologous bone flap are included in a clinical and image-based follow-up to identify cases and severity of bone flap resorption.

The explanted autologous bone flaps are cryoconserved and reimplanted at a time-point defined by the surgeon according to standards of the participating hospital. The fixation of the bone flap is also performed according to the surgeon's decision.

A cranial CT is performed within one week after reimplantation to define a baseline.

A second, only clinical, follow-up will take place within 2 months after reimplantation.

Two more follow-ups including photodocumentation of the cranial and facial symmetry (portrait and profile) and cranial CT will take place 12 and 24 months after reimplantation.

The indication for surgical revision in case of bone flap resorption is independent from the study and falls under the responsibility of the treating surgeon.

ELIGIBILITY:
Inclusion Criteria:

* all patients after hemicraniectomy or bifrontal craniectomy
* age 18-99 y/o
* ability to understand and sign informed consent (alternatively, legal representative may sign)

Exclusion Criteria:

* bone flap not fit for reimplantation
* no cryoconservation performed but other technique
* pregnancy
* patient's death

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing reimplantation of cryoconserved bone flaps after craniectomy
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-01; Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of a relevant bone resorption within 12 months after reimplantation | 12 months
  The extent of bone flap resorption is analyzed as well objectivela as subjectivels:
  objective criteria: Volumetric reconstruction of the bone flap from the CT scans and subtration of the actual bone flap volume from the 3D model at the basline-timepoint directly after reimplantation
  subjective: a bone flap resorption score is validated

SECONDARY OUTCOMES:
Incidence of an indication for surgical revision | 12 and 24 months after reimplantation
  The indication for a surgical revision falls under responsibility of the treating surgeon.
Death | 2, 12 and 24 months after reimplantation
  death
Infections | 2, 12 and 24 months after reimplantation
  Infections
Fluid collections and bleedings | 2, 12 and 24 months after reimplantation
  subgaleal, epidural and subdural fluid collections and hematomas
Hydrocephalus | 2, 12 and 24 months after reimplantation
  hydrocephalus
Temporal muscle atrophy | 2, 12 and 24 months after reimplantation
  temporal muscle atrophy
timepoint between explantation and reimplantation | 2, 12 and 24 months after reimplantation
  measured in months
patient age | 2, 12 and 24 months after reimplantation
  in years
fragmentation of the bone flap | 2, 12 and 24 months after reimplantation
  in number of pieces
temperature used for cryoconservation | 2, 12 and 24 months after reimplantation
  in °C
pathologies leading to explantation of the bone flap (hemicraniectomy) | 2, 12 and 24 months after reimplantation
  trauma, tumor, stroke and others

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern
  - Dept. of Neurosurgery, Zurich University Hospital, Zurich